CLINICAL TRIAL: NCT02509715
Title: Effect of Intraoperative Nerve Monitoring on Voice Quality During Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lütfiye Nuri Burat Government Hospital (Other Government)
Responsible Party: Principal Investigator, TURGUT DONMEZ, General Surgeon, MD, Lütfiye Nuri Burat Government Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEAH-2015-17
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Thyroid
Keywords: thyroidectomy; nerve monitoring
MeSH Terms: conditions — Thyroid Diseases | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Conventional group (No Intervention): Standard conventional thyroid surgery
- IONM group (Active Comparator): Intraoperative nerve monitoring used thyroid surgery
  Interventions: Procedure: Intraoperative nerve monitoring

INTERVENTIONS:
Procedure: Intraoperative nerve monitoring — Intraoperative nerve monitoring during thyroid surgery
  Arms: IONM group

SUMMARY:
"Effect of intraoperative nerve monitoring on voice quality during thyroid surgery"

Thyroidectomy is a quite often surgical procedure applied by both head and neck surgeons and endocrine surgeons.Recent advances in surgical and technological area achieve a remarkable decrease in the complication rates. In case of these advances, patients still have fear related with their voice. In this study, investigators aimed to investigate voice changes during thyroid surgery and effect of intraoperative nerve monitoring to the voice quality.

DETAILED DESCRIPTION:
In order to minimize the complication rates and voice disturbances during thyroidectomy, intraoperative nerve monitoring(IONM) is a widely used intervention. In this study investigators will compare conventional surgery with IONM used surgery. Randomly chosen half of the patients will be operated with IONM. Vagus, recurrent and superior laryngeal nerves will be monitored during surgery and measured for nerve integrity . Rest of the patients will be operated with standard conventional method. All participants will be analyzed with a computer program for their voice quality preoperatively and postoperatively at 14th day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of nodular or multinodular goiter
* Clinical, radiological and pathologically diagnosed thyroid cancer
* Must be able to speak (for voice recording)

Exclusion Criteria:

* Pregnancy
* Previous thyroid surgery
* Previous laryngeal operations
* Professional voice users (e.g. singers)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-09 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Voice analysis | up to 2nd week voice recording
  Comparison of Jitter(microseconds) and Shimmer(dB) values of recorded voices

SECONDARY OUTCOMES:
Operation time | duration of surgery, up to 3 hours
  Comparison of differences in operation time period between the groups whether IONM used or not

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, MD, Principal Investigator — Lutfiye Nuri Burat Goverment Hospital
Locations (1):
- Lutfiye NBGH, Istanbul, Turkey (Türkiye)